CLINICAL TRIAL: NCT03982589
Title: Telomere Length in Relation to Acute Stress Response in Critical Care Patients
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0319-11-RMC
Record Dates: First submitted 2019-06-10; First posted 2019-06-11 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Acute Disease; Telomere Shortening
MeSH Terms: conditions — Acute Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — telomere extracted from white blood cells (WBC) anonymously
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the investigators studied the impact of severe stress (in this case any event or illness leading to a necessity of critical care) on telomere length.

DETAILED DESCRIPTION:
Telomeres length analysis were determined from 2 blood samples, the initial sample drawn in the first 72 hours after hospitalization and the second after not < 5 or > 14 days. For patients discharged before day 5, a repeat sample was drawn and analyzed on the discharge day. The blood sample processing was as follows: 5 ml of blood was collected and the red blood cells (RBC) were lysed using the RBC lysis solution (Biological Industries, Beit Haemek, Israel). Isolation of genomic DNA was performed by using the DNA isolation kit for mammalian blood (Roche, Mannheim, Germany). Briefly, DNA was isolated by the salting out procedure, washed and precipitated by isopropanol. The DNA was resuspended in polymerase chain reaction (PCR) grade water. The DNA concentration was measured by using the NanoDrop device (Thermo Fisher, USA).

DNA samples were analyzed for telomere length according to the method of Cawthon (2009) [20] with slight modifications. Each DNA sample was analyzed by two sets of primers detailed below, one for telomere length analysis and one for a reference gene analysis (human hemoglobin). The primers were diluted to 100µM in PCR grade water and then to 10µM. DNA samples were diluted to 2.5 ng/µl in PCR grade water. The primers sequences are shown below:

telc: TGTTAGGTATCCCTATCCCTATCCCTATCCCTATCCCTAACA telg: ACACTAAGGTTTGGGTTTGGGTTTGGGTTTGGGTTAGTGT hbgd:_GCCCGGCCCGCCGCGCCCGTCCCGCCGGAGGAGAAGTCTGCCGTT hbgu: GGCGGCGGGCGGCGCGGGCTGGGCGGCTTCATCCACGTTCACCTTG

Reaction PCR were processed as follows:

50°C for 2 min, 95°C for 5 min, a single cycle of 94°C for 15 sec, 49°C for 15 sec; 40 cycles of: 94°C for 15sec, 62°C for 10 sec and a final stage of: 74°C for 15 sec. All reactions were performed using the Step One device (ABI, USA).

ELIGIBILITY:
Inclusion Criteria:

* • Patients hospitalized up to 72 hours prior to admission to the ICU

  * Predicted ICU stay is at least 5 days

Exclusion Criteria:

* • Pregnancy and lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults (male and females) admitted to the ICU
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
telomere length difference | 7 days
  the difference between telomere length in percent between samples taken

SECONDARY OUTCOMES:
correlation between mortality and telomere length | 6 month
  correlation between mortality and telomere length
correlation between telomere length change and leukocytes count change | 7 days
  correlation between telomere length change and leukocytes count change

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin medical center, Petah Tikva, Israel